CLINICAL TRIAL: NCT00219453
Title: A Pilot Safety Study to Determine the Presence of Hepatitis B Virus in Downstream Injection Samples Using the HSI-500 Jet Injector With Protector Cap
Brief Title: Pilot Safety Study to Determine the Ability of the Protector Cap Jet Injector to Prevent Cross-Contamination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS243
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Virus Diseases; Hepatitis B
Keywords: Pilot Projects; Injections, Jet; Injections, Jet/instrumentation; Equipment Contamination/prevention and control; Blood-Borne Pathogens; Disease Transmission, Horizontal
MeSH Terms: conditions — Virus Diseases; Hepatitis B

INTERVENTIONS:
Device: Jet Injector with Protector Cap (HSI-500)

SUMMARY:
The primary purpose of this study is to determine the ability of the Protector Cap Jet Injector to prevent cross-contamination in the next injection sample. The hypothesis is that the Protector Cap Jet Injector will prevent contamination in the next injection sample, even following injection of volunteers with high levels of hepatitis B virus.

DETAILED DESCRIPTION:
The jet injector is a needle-free injection device that uses a high-pressure stream to penetrate the skin and deliver medication into intradermal, subcutaneous, or intramuscular tissues. Multi-dose jet injectors are a type of jet injector with a reusable fluid path that consists of the vial adapter, dose chamber, fluid pathway, and nozzle. Although credited with decades of use and the delivery of millions of doses of vaccine in the field, multi-dose jet injectors are no longer used due to evidence of cross-contamination between injections. The HSI-500 Jet Injector with Protector Cap has been designed with a disposable plastic cap that acts as a shield between the nozzle and the skin to eliminate cross-contamination between injections while maintaining a high rate of vaccine delivery to multiple patients.

The objective of this pilot safety study is to provide a preliminary indication of the ability of the jet injector to prevent cross-contamination from hepatitis B virus between volunteer injections. A secondary objective of the study is to test study procedures prior to a larger-scale safety study.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18 and 60 years.
* Either male or female.
* In good health, by self-report and confirmed by physical exam.
* Willing and able to follow procedural requirements of the study.
* Willing and able to provide informed consent for study participation.
* Ability to read and understand informed consent information sheet in English.

For Hepatitis B Positive Volunteers

* Actively infected with blood levels of greater than or equal to 10*6 hepatits B virus (HBV) copies/mL, confirmed by HBV DNA blood test conducted up to 21 days prior to the day of study enrollment (existing patient record)
* Not presently taking any heparin-based drugs that could potentially interfere with HBV assays.

For Hepatitis B Negative Volunteers

* Not actively infected with HBV as confirmed by HBV tests.
* Not presently taking any drugs that could potentially interfere with HBV assays.
* No prior history of HBV infection.

Exclusion Criteria:

* Requires anti-viral HBV therapy.
* History of allergic reactions or anaphylaxis to immunizations.
* Dermatological conditions affecting the injection site (such as eczema).
* Blood coagulation disorders or history of taking drugs that affect blood coagulation.
* Presently taking any heparin-based medication (Calciparine, Liquaemin Sodium, Hep-Lock, or Hep-Lock U/P) that could potentially interfere with HBV assays.
* History of severe psychiatric disease.
* Previous suicidal attempt or hospitalization for psychiatric episode within the last 24 weeks.
* Any other conditions or circumstances that, in the opinion of the investigator, may be a threat to the safety and welfare of the volunteer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17
Dates: Start 2004-10; Study Completion 2006-01

PRIMARY OUTCOMES:
Presence of hepatitis B virus in post-injection saline samples as verified by a polymerase chain reaction (PCR)-based assay

SECONDARY OUTCOMES:
Evaluation of injection site reactions by observation and self-report of pain on a scale (none, mild, moderate, severe)

CONTACTS AND LOCATIONS:
Overall Officials: Darin L Zehrung, BS, Study Director — PATH

REFERENCES:
- See also: August 9, 2005 FDA Safety Panel meeting information: agenda, meeting transcript, questions, and other supporting documentation. — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfAdvisory/details.cfm?mtg=556